## INFORMED CONSENT

Fitforlife; Peer-mentor driven physical exercise for persons affected by psychosis.

1.6.2019

## **FitForLife**

## **Informed consent**

I have received information about the Fitforlife study and have been able to discuss and hereby agree to participate. I agree to that personal data are saved and that my blood samples will be saved in a biobank.

I am aware that I can withdraw at any time and that this will not affect my usual care.

Signature, Name and Date